CLINICAL TRIAL: NCT05179590
Title: Factors Associated With Quality of Dreams During General Anesthesia: a Prospective Observational Study
Brief Title: Factors Associated With Quality of Dreams During General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Bijia Song, principal investigator, Beijing Friendship Hospital
Other Study IDs: General anesthesia and dream
Record Dates: First submitted 2021-12-17; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Dream; General Anesthesia; Perioperative Factors; Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General anesthesia Group
  Interventions: Other: Quality of Dream

INTERVENTIONS:
Other: Quality of Dream — Patients frequently report having dreams during general anesthesia, and the dreams are often reported to be pleasant dreams.
  However, factors associated with the quality of dreams during general anesthesia have not been clarifed. The aim of this study was to determine the relationships between the quality of dreams during general anesthesia and perioperative factors.
  This prospective observational study included patients scheduled for elective surgery under general anesthesia.

SUMMARY:
Patients frequently report having dreams during general anesthesia. The incidence of dreams during general anesthesia that have been reported by patients upon awakening has been reported to range from 10 to 36% [1] and to be higher in younger patients, female patients [2], and patients who received ketamine [3]. The quality of dreams during general anesthesia is often reported as pleasant, but some patients report unpleasant or not pleasant dreams [4, 5]. However, the factors associated with the quality of dreams have remained to be elucidated. Therefore, the aim of this study was to determine the relationships between the quality of dreams during general anesthesia and perioperative factors.

ELIGIBILITY:
Inclusion Criteria:

* We recruited patients who were more than 20 years of age
* Patients who were scheduled for elective surgery under general anesthesia regardless of the type of surgery

Exclusion Criteria:

* diagnosis of a psychological disorder,
* major afective disorder
* major drug dependence disorder,
* inability to understand the content of our study,
* planned postoperative ventilation,
* anticipation of unavailability for postoperative interviews

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We recruited patients who were more than 20 years of age and who were scheduled for elective surgery under general anesthesia regardless of the type of surgery
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Anesthesia information | During the operation
  Anesthesia was maintained with a general anesthetic (propofol, sevofurane, or desfurane) and remifentanil. Some patients also received a peripheral nerve block. Anesthetic management including the choice of a general anesthestic (propofol, sevofurane, or desflurane) depended on the decision of the anesthesiologists in charge
Dream interview | After extubation, patients were interviewed about intraoperative dreams in the operating room as soon as they were oriented to time, place, and person
  The following questions were asked.
  1. What was the last thing you remember before going to sleep?
  2. What was the frst thing you remember from when you woke up?
  3. Can you recall anything between?
  4. Did you have any dreams while under anesthesia?
  5. How did you feel about your dream: pleasant, indiferent or unpleasant?
Depression level | the day before surgery
  The Hospital Anxiety and Depression Scale (HADS), which is a self-report questionnaire, was used for evaluation of anxious and depressive states in the participants